CLINICAL TRIAL: NCT02121262
Title: Dexamethasone Posterior Segment Drug Delivery System Versus Laser Photocoagulation in Patients With Diabetic Macular Edema
Brief Title: A Safety and Efficacy Study of Dexamethasone Versus Laser Photocoagulation in Participants With Diabetic Macular Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206207-026
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Photocoagulation (Other): Laser photocoagulation was administered in the study eye on Day 1, and on Months 3, 6, and 9, if retreatment indicated.
  Interventions: Procedure: Laser Photocoagulation
- Dexamethasone (Experimental): Dexamethasone 700 μg was administered as intravitreal injection in the study eye on Day 1, Months 5, and 10.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 700 μg intravitreal injection in the study eye on Day 1, Months 5, and 10.
  Other Names: OZURDEX®
  Arms: Dexamethasone
Procedure: Laser Photocoagulation — Laser photocoagulation on Day 1, and on Months 3, 6, and 9, if retreatment indicated.
  Arms: Laser Photocoagulation

SUMMARY:
This study will evaluate the safety and efficacy of 700 μg dexamethasone versus laser photocoagulation in participants with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2)
* Presence of macular edema

Exclusion Criteria:

* Anticipated need for ocular surgery in the study eye during the study
* Laser photocoagulation in the study eye within 3 months
* Cataract surgery within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Li, Study Director — Allergan
Locations (18):
- China (16):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - People's Hospital of Peking University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing TongRen Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Zhongshan Ophthalmic Center, Sun Yet-Sen University, Guangzhou, Guangdong
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The 2nd hospital of JiLin University, Changchun, Jilin
  - The Eye and ENT Hospital, Affiliated of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - TianJin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Wenzhou Ophthalmic Centre, Wenzhou, Zhejiang
- Philippines (2):
  - Asian Eye Institute, Makati City, National Capital Region
  - Peregrine Eye and Laser Institute, Makati City, National Capital Region

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Photocoagulation | Dexamethasone
Started | 139 | 145
Treated | 129 | 145
Modified Intent-to-treat Population | 127 | 145
Completed | 108 | 135
Not Completed | 31 | 10
Not completed — Adverse Event | 6 | 3
Not completed — Lack of Efficacy | 3 | 0
Not completed — Personal Reasons | 19 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Participant Dropped-out | 0 | 1
Not completed — Participant was Deemed Unsuitable | 1 | 0
Not completed — Consent Withdrawn | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) population included all randomized and treated participants with at least one postbaseline best corrected visual acuity (BCVA) measurement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser Photocoagulation | Dexamethasone | Total
Number analyzed (Participants) | 127 | 145 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (7.73) | 59.1 (8.08) | 59.3 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 64 | 133
  Male | 58 | 81 | 139
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 127 | 145 | 272
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 113 | 129 | 242
  Ethnicity: Other | 14 | 16 | 30
BCVA in the Study Eye [Mean (Standard Deviation); unit: letters] — BCVA was measured using an eye chart and is reported as the number of letters read correctly using the early treatment diabetic retinopathy study (ETDRS) scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The eligible eye with worse visual acuity was selected as the study eye.
  letters | 55.1 (10.32) | 55.7 (11.44) | 55.4 (10.91)
Central Retinal Thickness (CRT) by Optical Coherence Tomography (OCT) in the Study Eye [Mean (Standard Deviation); unit: microns] — CRT was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system that provides high-resolution imaging sections of the retina. SD-OCT is performed in the study eye after pupil dilation. The eligible eye with worse visual acuity was selected as the study eye.
  microns | 482.1 (154.39) | 491.2 (160.80) | 486.9 (157.61)
Total Macular Leakage Area by Fluorescein Angiography (FA) in the Study Eye [Mean (Full Range); unit: mm^2] — FA is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Early and transit images were taken of the study eye. Mid- and late-phase images were taken of the study eye and non-study eye. Electronic FA images were collected for evaluation by a reading center to identify macular area of leakage. The eligible eye with worse visual acuity was selected as the study eye. Population: Data for Total Macular Leakage Area was only available for 125 participants in the Laser Photocoagulation arm.
  mm^2 | 30.076 [2.81 to 40.78] | 29.644 [1.69 to 40.71] | 29.8 [1.69 to 40.78]

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With BCVA Improvement ≥15 Letters From Baseline in the Study Eye
Description: BCVA was measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The eligible eye with worse visual acuity was selected as the study eye.
Time Frame: Baseline to Month 12
Population: mITT population included all randomized and treated participants with at least one postbaseline BCVA measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Laser Photocoagulation | Dexamethasone
Number analyzed (Participants) | 127 | 145
percentage of participants | 10.2 | 11.7
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Dexamethasone; Test type: Superiority; p = 0.7431, Cochran-Mantel-Haenszel; Based on the Cochran-Mantel-Haenszel (CMH) general association test stratified by baseline BCVA categories; Rate Difference = 1.5, 95% CI 2-sided [-5.9 to 8.9]

2. Primary Outcome: Average Change From Baseline (CFB) in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA was measured using an eye chart and is reported as the number of letters read correctly using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. The eligible eye with worse visual acuity was selected as the study eye. The average change was computed by subtracting the baseline BCVA from the area under the BCVA curve (AUC) divided by the total follow-up time for each participant. Analysis of covariance (ANCOVA) model was used for the analysis.
Time Frame: Baseline to Month 12
Population: mITT population included all randomized and treated participants with at least one postbaseline BCVA measurement.
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | Laser Photocoagulation | Dexamethasone
Number analyzed (Participants) | 127 | 145
letters | 1.4 (0.65) | 4.3 (0.61)
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Dexamethasone; Test type: Superiority; p = 0.0011, ANCOVA; The ANCOVA model included the treatment group as the main effect and baseline BCVA score as the covariate; Least Squares Mean (LSM) Difference = 2.9, 95% CI 2-sided [1.17 to 4.66], Standard Error of Mean 0.89 — Null hypothesis-there was no difference in treatment groups of average BCVA CFB in 12-months. Hypothesis test-based on 2-sided test at 0.05 significance level,confidence interval(CI) was constructed between treatment groups in LSM using ANCOVA model

3. Secondary Outcome: Change From Baseline in CRT by Spectral Domain Optical Coherence Tomography (SD-OCT) in the Study Eye
Description: CRT was assessed using SD-OCT, a non-invasive diagnostic system that provides high-resolution imaging sections of the retina. SD-OCT is performed in the study eye after pupil dilation. A negative change from Baseline indicates improvement and a positive change from baseline indicates worsening. The eligible eye with worse visual acuity was selected as the study eye. ANCOVA model was used for the analysis.
Time Frame: Baseline to Month 12
Population: mITT population included all randomized and treated participants with at least one postbaseline BCVA measurement. Last observation carried forward (LOCF) was used
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | Laser Photocoagulation | Dexamethasone
Number analyzed (Participants) | 127 | 145
microns | -120.3 (13.20) | -209.5 (12.27)
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Dexamethasone; Test type: Superiority; p < 0.0001, ANCOVA; Based on ANCOVA model with treatment and baseline BCVA categories as main effects and baseline retinal thickness as the covariate; Least Squares Mean Difference = -89.3, 95% CI 2-sided [-122.53 to -56.01], Standard Error of Mean 16.89 — Null hypothesis was there was no difference in treatment groups in average BCVA CFB in 12-months. Hypothesis test was based on 2-sided test at 0.05 significance level. 2-sided 95% CI was constructed between treatment groups in LSM using ANCOVA model

4. Secondary Outcome: Change From Baseline in Total Macular Leakage Area by FA in the Study Eye
Description: FA is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Early and transit images were taken of the study eye. Mid- and late-phase images were taken of the study and non-study eye. Electronic FA images were collected for evaluation by a reading center. The eligible eye with worse visual acuity was selected as the study eye. ANCOVA model was used for the analysis.
Time Frame: Baseline to Month 12
Population: mITT population included all randomized and treated participants with at least one postbaseline BCVA measurement. LOCF was used. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Laser Photocoagulation | Dexamethasone
Number analyzed (Participants) | 125 | 145
mm^2 | -0.637 (0.8133) | -8.367 (0.7482)
Statistical Analysis 1: Comparison: Laser Photocoagulation vs Dexamethasone; Test type: Superiority; p < 0.0001, ANCOVA; Based on ANCOVA model with treatment and baseline BCVA categories as main effects and baseline total leakage area as the covariate; Least Squares Mean Difference = -7.729, 95% CI 2-sided [-9.7855 to -5.6733], Standard Error of Mean 1.0443 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first dose up to last dose (Up to Month 12)
Description: Safety Population included all participants who received the study medication or had the study procedure performed on the study eye.
Arm/Group | Laser Photocoagulation | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/129 | 2/145
Serious Adverse Events (participants affected / at risk) | 21/129 | 35/145
Other Adverse Events (participants affected / at risk) | 51/129 | 99/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Photocoagulation (N=129) | Dexamethasone (N=145)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 4
Coronary artery disease (Cardiac disorders) | 4 | 2
Myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 8
Vitreous haemorrhage (Eye disorders) | 1 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Photocoagulation (N=129) | Dexamethasone (N=145)
Cataract (Eye disorders) | 8 | 16
Visual impairment (Eye disorders) | 18 | 15
Ocular hypertension (Eye disorders) | 1 | 10
Dry eye (Eye disorders) | 7 | 8
Vitreous haemorrhage (Eye disorders) | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 13
Conjunctivitis (Infections and infestations) | 2 | 13
Nasopharyngitis (Infections and infestations) | 4 | 8
Urinary tract infection (Infections and infestations) | 8 | 4
Intraocular pressure increased (Investigations) | 9 | 50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT02121262/SAP_000.pdf
  • Study Protocol (2013-04-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT02121262/Prot_001.pdf